CLINICAL TRIAL: NCT01933152
Title: Review Study: A Retrospective Noninterventional Study to Assess the EffectiVeness of exIsting Anti-vascular Endothelial groWth Factor (Anti-VEGF) Treatment Regimens in Patients With Wet Age-related Macular Degeneration
Brief Title: Study to Assess the EffectiVeness of exIsting Anti-vascular Endothelial groWth Factor (Anti-VEGF) Treatment Regimens in Patients With Wet Age-related Macular Degeneration
Acronym: REVIEW
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 16378
Record Dates: First submitted 2013-07-29; First posted 2013-09-02 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Macular Degeneration
Keywords: wAMD; anti-VEGF
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — Patients with wet AMD treated with ranibizumab as prescribed by physician

SUMMARY:
Retrospective, non-interventional, observational multi-center field study. Patients diagnosed with wet Age-related macular degeneration (wAMD) and having started treatment with ranibizumab between January 1, 2009 and December 31, 2009 must be consecutively screened and, if eligible, enrolled. Patients will be followed up at maximum until December 31, 2011. Switch to any other Anti vascular endothelial growth factor (anti VEGF) treatment will be documented. For each patient, demographics, medical history, administered treatments, results of ocular and visual assessments and other tests (where available) will be documented.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of wet Age-related Macular Degeneration
* Start of anti-VEGF therapy with ranibizumab (Lucentis) between January 1, 2009 and December 31, 2009
* Informed consent form signed

Exclusion Criteria:

- Participation in an investigational study during anti-VEGF therapy (from start up to December 31, 2011) that involved treatment with any drug or device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients must have been diagnosed to suffer from wet AMD and must have started anti-VEGF treatment with ranibizumab between January 1, 2009, and December 31, 2009
Sampling Method: Non-Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2012-08; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Changes in visual acuity after start of Anti vascular endothelial growth factor (anti VEGF) therapy with ranibizumab, assessed by Early Treatment Diabetic Retinopathy (ETDRS) or Snellen chard | Baseline and 24 months

SECONDARY OUTCOMES:
Demographic characteristics of patients included in the study (Age, Sex, Race) | Baseline
Mean time from first clinical presentation to diagnosis | Baseline
Mean time from diagnosis to treatment | Time from diagnosis to treatment: Up to 24 months
Mean time from diagnosis to end of follow-up | Time from diagnosis to end of follow-up: up to 48 months
Mean change of visual acuity, from diagnosis to end of follow-up, assessed by Early Treatment Diabetic Retinopathy (ETDRS) or Snellen chart | Baseline and 24 months
Mean change of retinal thickness from diagnosis to end of follow-up, assessed by Optical Coherence Tomography (OCT) | Baseline and 24 months
Mean change of lesion size from diagnosis to end of follow-up, assessed by Fluorescein Angiography (FA) | Baseline and 24 months
Average number of treatments given from diagnosis to end of follow-up | After 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Portugal